CLINICAL TRIAL: NCT01804465
Title: A Randomized Phase 2 Trial of Immediate vs. Delayed Anti-CTLA4 Blockade Following Sipuleucel-T Treatment for Prostate Cancer Immunotherapy
Brief Title: Sipuleucel-T With Immediate vs. Delayed Cytotoxic T-Lymphocyte-Associated Protein 4 (CTLA-4) Blockade for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Bristol-Myers Squibb (Industry); Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12557; NCI-2014-00318 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2013-02-27; First posted 2013-03-05 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
Keywords: castration resistant; prostate; cancer; ipilimumab; provenge; SipT
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — sipuleucel-T; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate IpilimumabTreatment (Experimental): Arm 1 (Immediate Treatment) Ipilimumab Q3wks x 4 started 1 day following the final dose of SipT.
  Interventions: Drug: SipT Treatment; Drug: Ipilimumab
- Delayed IpilimumabTreatment (Experimental): Arm 2 (Delayed Treatment) Ipilimumab Q3wks x 4 started 3 weeks following the final dose of SipT.
  Interventions: Drug: SipT Treatment; Drug: Ipilimumab

INTERVENTIONS:
Drug: SipT Treatment — All patients will receive standard of care SipT treatment every two weeks for a total of 3 treatments. The three treatments usually take about 30 days to complete.
  SipT treatment is given in three 1 hour infusions. Each SipT treatment is generated from a standard blood cell-collection procedure (called leukapheresis) performed 2-3 days prior to the infusion.
  Other Names: Provenge
Drug: Ipilimumab — Ipilimumab will be given by IV over 90 minutes every 3 weeks. Patients will be monitored during the infusion and up to 1 hour post-infusion.
  Other Names: BMS-734016/MDX-010, anti-CTLA4

SUMMARY:
The purpose of this study is to find out what effects taking ipilimumab, as an immediate or delayed treatment, following completion of sipuleucel-T (SipT) treatment, has on patients and their prostate cancer.

DETAILED DESCRIPTION:
This is an open-label randomized multicenter Phase 2 clinical trial combining SipT with ipilimumab in patients with chemotherapy-naïve metastatic castration resistant prostate cancer (CRPC).

All patients will be treated with standard SipT (Q2wks x 3). Patients will be randomized to one of two arms:

Arm 1 (Immediate Treatment): Ipilimumab Q3wks x 4 started 1 day following the final dose of SipT (Day 0).

Arm 2 (Delayed Treatment): Ipilimumab Q3wks x 4 started 3 weeks following the final dose of SipT (Day 0).

Following this ipilimumab treatment, patients will then be followed monthly for 3 months and then quarterly until disease progression. The definition of unacceptable toxicity is grade 3 or higher treatment-related toxicities (NCI CTCAE v4) excluding immune-related adverse events (irAEs). The study will assess for the immunogenicity and clinical activity of sequential sipuleucel-T treatment followed by ipilimumab. Patients who experience an initial clinical response to ipilimumab followed by subsequent disease progression will be offered reinduction treatment with ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, metastatic prostate adenocarcinoma (positive bone scan and/or measurable disease on CT scan and/or MRI of the abdomen and pelvis).
2. Progressive disease after androgen deprivation, as defined by Prostate Cancer Clinical Trials Working Group 2 (PCWG2) and/or RECIST criteria. Patients must have disease progression by one or both of the following:

   * For patients with measurable disease, progression is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions or the appearance of one or more new lesions, as per RECIST criteria version 1.1.
   * For patients with no measurable disease, a positive bone scan and elevated prostate specific antigen (PSA) will be required. PSA evidence for progressive prostate cancer consists of a PSA level of at least 2 ng/milliliter (mL), which has risen on at least 2 successive occasions, at least 1 week apart. If the confirmatory PSA value is not greater than the screening PSA value, then an additional test for rising PSA will be required to document progression.
   * If no prior orchiectomy has been performed, patients must remain on luteinizing hormone-releasing hormone (LHRH) agonist or antagonist (e.g. degarelix) therapy. Patients who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of the antiandrogen, defined as two consecutive rising PSA values, obtained at least two weeks apart, or documented osseous or soft tissue progression. At least one of the PSA values must be obtained at least four weeks (flutamide) or six weeks (bicalutamide or nilutamide) after discontinuation.
3. Laboratory requirements:

   * Absolute neutrophil count (ANC) ≥ 1500/μL
   * Bilirubin < 1.5 x upper limit of normal (ULN)
   * Hemoglobin ≥ 8 g/dL
   * PSA ≥ 2 ng/mL
   * Platelets ≥ 100,000/μL
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x ULN
   * Creatinine clearance ≥ 60 mL/min by the Cockcroft Gault equation
   * Testosterone less than or equal to 50 ng/dL
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1 and life expectancy ≥ 12 weeks.
5. At least 18 years of age or older.
6. Patients receiving any other hormonal therapy, including any dose of megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g. Saw Palmetto, PC-SPES), or any systemic corticosteroid, must discontinue the agent for at least four weeks prior to study treatment. Progressive disease as defined above must be documented after discontinuation of any hormonal therapy (with the exception of a LHRH agonist).
7. Prior radiation therapy must be completed ≥ 4 weeks prior to enrollment and the patient must have recovered from all toxicity. Prior radiopharmaceuticals (strontium, samarium) must be completed ≥ 8 weeks prior to enrollment.
8. Because of the unknown potential risk to a gamete and/or developing embryo from these investigational therapies, patients must agree to use adequate contraception (barrier method for males) for the duration of study participation, and for three months after discontinuing therapy.

Exclusion Criteria:

1. Prior chemotherapy for prostate cancer, with the exception of neoadjuvant chemotherapy, because of the potential effect of chemotherapy on the immune system.
2. Prior sipuleucel-T treatment or investigational immunotherapy.
3. Prostate cancer pain requiring regularly scheduled narcotics.
4. Current treatment with systemic steroid therapy (inhaled/topical steroids are acceptable). Systemic corticosteroids must be discontinued for at least 4 weeks prior to first treatment.
5. History of autoimmune disease including, but not limited to:

   * Systemic lupus erythematosis (SLE), scleroderma, CREST syndrome, rheumatoid arthritis
   * Inflammatory bowel disease, celiac disease, primary biliary cirrhosis, autoimmune hepatitis
   * Dermatomyositis, polymyositis, giant cell arteritis
   * Autoimmune hemolytic anemia (AIHA), cryoglobulinemia, antiphospholipid antibody syndrome (APLS)
   * Diabetes mellitus type I, myasthenia gravis, Grave's disease
   * Wegener's granulomatosis or other vasculitis
   * A history of Hashimoto's thyroiditis, psoriasis, or eczema, any of which has been inactive for at least one year, or isolated Raynaud's phenomenon is acceptable
6. Known central nervous system or visceral metastases.
7. Medical or psychiatric illness that would, in the opinion of the investigator, preclude participation in the study or the ability of patients to provide informed consent for themselves.
8. Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association Class III or IV), active angina pectoris, or recent myocardial infarction (within the last 6 months).
9. Concurrent or prior malignancy except for the following:

   * Adequately treated basal or squamous cell skin cancer
   * Adequately treated stage I or II cancer from which the patient is currently in complete remission
   * Any other cancer from which the patient has been disease-free for 5 years
10. Known HIV or other history of immunodeficiency disorder.
11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or medical (e.g. infectious) illness.
12. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of adverse events (AE), such as a condition associated with frequent diarrhea.
13. A history of prior treatment with ipilimumab or prior cluster of differentiation 137 (CD137) agonist or CTLA-4 inhibitor or agonist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, MD, Principal Investigator — University of California, San Francisco; Padmanee Sharma, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sinha M, Zhang L, Subudhi S, Chen B, Marquez J, Liu EV, Allaire K, Cheung A, Ng S, Nguyen C, Friedlander TW, Aggarwal R, Spitzer M, Allison JP, Small EJ, Sharma P, Fong L. Pre-existing immune status associated with response to combination of sipuleucel-T and ipilimumab in patients with metastatic castration-resistant prostate cancer. J Immunother Cancer. 2021 May;9(5):e002254. doi: 10.1136/jitc-2020-002254. PMID 33986125

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate IpilimumabTreatment: Arm 1 (Immediate Treatment) Ipilimumab Q3wks x 4 started 1 day following the final dose of Sipuleucel-T (SipT).
  SipT Treatment: All patients will receive standard of care SipT treatment every two weeks for a total of 3 treatments. The three treatments usually take about 30 days to complete.
  SipT treatment is given in three 1 hour infusions. Each SipT treatment is generated from a standard blood cell-collection procedure (called leukapheresis) performed 2-3 days prior to the infusion.
  Ipilimumab: Ipilimumab will be given by IV over 90 minutes every 3 weeks. Patients will be monitored during the infusion and up to 1 hour post-infusion.
- Delayed IpilimumabTreatment: Arm 2 (Delayed Treatment) Ipilimumab Q3wks x 4 started 3 weeks following the final dose of SipT.
  SipT Treatment: All patients will receive standard of care SipT treatment every two weeks for a total of 3 treatments. The three treatments usually take about 30 days to complete.
  SipT treatment is given in three 1 hour infusions. Each SipT treatment is generated from a standard blood cell-collection procedure (called leukapheresis) performed 2-3 days prior to the infusion.
  Ipilimumab: Ipilimumab will be given by IV over 90 minutes every 3 weeks. Patients will be monitored during the infusion and up to 1 hour post-infusion.
Period: Overall Study
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Immediate IpilimumabTreatment: Arm 1 (Immediate Treatment) Ipilimumab Q3wks x 4 started 1 day following the final dose of SipT.
  SipT Treatment: All patients will receive standard of care SipT treatment every two weeks for a total of 3 treatments. The three treatments usually take about 30 days to complete.
  SipT treatment is given in three 1 hour infusions. Each SipT treatment is generated from a standard blood cell-collection procedure (called leukapheresis) performed 2-3 days prior to the infusion.
  Ipilimumab: Ipilimumab will be given by IV over 90 minutes every 3 weeks. Patients will be monitored during the infusion and up to 1 hour post-infusion.
- Total: Total of all reporting groups
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 3 | 2 | 5
  60-69 years old | 13 | 15 | 28
  70-79 years old | 8 | 9 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 26 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 17 | 23 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Immune Response to Prostatic Acid Phosphatase (PAP) and/or PA2024
Description: Immune response will be tested using the single sample binomial exact test when induction therapy is completed. The Immunoglobulin M (IgM) and Immunoglobulin G (IgG) antibody responses to PAP and/or PA2024 will be assessed by ELISA assay at baseline and week 20 after start of sipT treatment (day 113 of study treatment). A positive response is defined as a titer > 1:400. The positive immune percentage for both IgG and IgM antibodies to PAP and to PA2024 will be used to summarize the results for each study arm.
Time Frame: Up to 20 weeks
Population: Only a small portion of the collected samples contained enough aliquots or tissue available for this particular analysis
Measure: Number; unit: percentage of participants
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 7 | 8
percentage of participants | 71.4 | 87.5

2. Primary Outcome: Proportion of Participants With Highest Grade, Treatment-related, Immune Response Adverse Events (IRAEs)
Description: Immune Response Adverse Events (IRAEs) will be reported for each study arm by tabulating the frequency of the maximum grade occurring for each patient for each type of iRAE using NCI Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0. IRAEs will be reported as a proportion of the participants in the treatment arm with the associated highest grade IRAE occurrences during protocol therapy.
Time Frame: Up to 20 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 24 | 26
proportion of participants
  Grade 2 Adrenal Insufficiency | 0.042 | 0.038
  Grade 3 Adrenal insufficiency | 0 | 0.038
  Grade 3 Diarrhea | 0.042 | 0.115
  Grade 4 Diarrhea | 0 | 0.038
  Grade 2 Hyperthyroidism | 0 | 0.038
  Grade 1 Hypothyroidism | 0 | 0.038
  Grade 2 Hypothyroidism | 0.042 | 0
  Grade 3 Lipase increased | 0.083 | 0.038
  Grade 2 Rash | 0.083 | 0.038
  Grade 3 Rash | 0.042 | 0

3. Secondary Outcome: Proportion of Patients Achieving a Prostate-specific Antigen (PSA) Decline of at Least 30% Below Baseline
Description: Descriptive statistics will be calculated to characterize the proportion of patients achieving a PSA decline of at least >30% after 1 cycle of treatment and presented along with the 95% confidence intervals for each study arm.
Time Frame: Up to 3 weeks
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 24 | 26
proportion | 0.125 [0.026 to 0.324] | 0.115 [0.025 to 0.302]

4. Secondary Outcome: Proportion of Patients Achieving a PSA Decline of at Least 50% Below Baseline
Description: Descriptive statistics will be calculated to characterize the proportion of patients achieving a PSA decline of at least >50% and presented along with the 95% confidence intervals for each study arm.
Time Frame: Up to 3 weeks
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 24 | 26
proportion | 0.083 [0.01 to 0.27] | 0.115 [0.025 to 0.302]

5. Secondary Outcome: Proportion of Patients Achieving an Objective Response
Description: Proportion of patients achieving an objective response as defined by Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) as complete response (irCR), partial response (irPR) will be reported along with 95% confidence intervals
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 24 | 26
proportion | 0 [NA to NA] — No participants achieved an objective response so a confidence interval could not be calculated | 0 [NA to NA] — No participants achieved an objective response so a confidence interval could not be calculated

6. Secondary Outcome: Proportion of Patients Achieving an Objective Response Stratified by Prior Radical Prostatectomy (RP)
Description: Proportion of patients achieving an objective response as defined by irRECIST as irCR +irPR and stratified by history of prior RP will be reported along with 95% confidence intervals.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 24 | 26
proportion | 0 [NA to NA] — No participants achieved an objective response so a confidence interval could not be calculated | 0 [NA to NA] — No participants achieved an objective response so a confidence interval could not be calculated

7. Secondary Outcome: Proportion of Patients Achieving an Objective Response Stratified by Radiation Therapy (RT)
Description: Proportion of patients achieving an objective response as defined by irRECIST as irCR + irPR stratified by prior RT will be reported along with 95% confidence intervals
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 24 | 26
proportion | 0 [NA to NA] — No participants achieved an objective response so a confidence interval could not be calculated | 0 [NA to NA] — No participants achieved an objective response so a confidence interval could not be calculated

8. Secondary Outcome: Radiographic Clinical Response Rate
Description: For each treatment arm, for patients with objective disease, using immune-related response criteria (irRC) criteria, the proportion of patients achieving a complete or partial response will be determined and reported with 95% confidence intervals
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 24 | 26
proportion | 0.833 [0.626 to 0.953] | 0.769 [0.564 to 0.91]

9. Secondary Outcome: Median Time to PSA Progression
Description: Time to PSA progression is defined as the start of protocol therapy to progression status at the end of 4 cycles of treatment as determined by the irRECIST.
Time Frame: Up to 12 weeks
Measure: Median (Full Range); unit: days
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
Number analyzed (Participants) | 24 | 26
days | 49 [-103 to 1092] | 47.5 [-54 to 414]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Immediate IpilimumabTreatment | Delayed IpilimumabTreatment
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/26
Serious Adverse Events (participants affected / at risk) | 1/24 | 11/26
Other Adverse Events (participants affected / at risk) | 21/24 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate IpilimumabTreatment (N=24) | Delayed IpilimumabTreatment (N=26)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Vascular Disorders - Other (Vascular disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate IpilimumabTreatment (N=24) | Delayed IpilimumabTreatment (N=26)
Diarrhea (Gastrointestinal disorders) | 4 (14) | 11 (19)
Nausea (Gastrointestinal disorders) | 3 (4) | 8 (13)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (9)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (6)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 8 (8) | 11 (20)
Pain (General disorders) | 8 (13) | 6 (14)
Fever (General disorders) | 5 (5) | 1 (2)
Chills (General disorders) | 0 (0) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (13)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Lipase increased (Investigations) | 5 (5) | 4 (7)
Investigations - Other (Investigations) | 2 (2) | 5 (8)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 3 (7)
Lymphocyte count decreased (Investigations) | 2 (4) | 2 (2)
Serum amylase increased (Investigations) | 3 (3) | 1 (1)
Weight loss (Investigations) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (5)
Alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 4 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 4 (4) | 3 (3)
Hematuria (Renal and urinary disorders) | 4 (5) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 3 (3) | 4 (6)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 3 (5)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (6) | 5 (7)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (5)
Upper respiratory infection (Infections and infestations) | 3 (3) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 3 (3)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT01804465/Prot_SAP_000.pdf